CLINICAL TRIAL: NCT02068027
Title: A Multicenter Randomized, Double-Blind, Placebo-Controlled, 2-Arm Parallel-Group Study to Determine the Efficacy and Safety of Clonidine Hydrochloride Topical Gel, 0.1% in the Treatment of Pain Associated With Painful Diabetic Neuropathy
Brief Title: Study of Clonidine Hydrochloride Topical Gel, 0.1% in the Treatment of Pain Associated With Diabetic Neuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioDelivery Sciences International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLO-290
Record Dates: First submitted 2014-02-19; First posted 2014-02-20 (Estimated); Results first posted 2017-08-24 (Actual); Last update posted 2017-09-26 (Actual); Status verified 2017-08

CONDITIONS: Painful Diabetic Neuropathy; Diabetic Neuropathy; Neuropathy
Keywords: Diabetes Mellitus; Pain; Foot pain; Neuropathy
MeSH Terms: conditions — Diabetic Neuropathies; Diabetes Mellitus; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clonidine Gel 0.1% (Experimental): Clonidine hydrochloride topical gel, 0.1%
  Interventions: Drug: Clonidine Gel 0.1%
- Placebo (Placebo Comparator): Placebo gel of identical appearance as active treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Clonidine Gel 0.1%
  Arms: Clonidine Gel 0.1%
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine whether clonidine gel is an effective treatment for reducing the pain associated with painful diabetic neuropathy.

DETAILED DESCRIPTION:
Study CLO 290 was a multicenter, randomized, double blind, placebo controlled, 2 arm parallel group study of Clonidine Gel in the treatment of pain associated with PDN. Subjects were randomly assigned in a 1:1 ratio to receive 1 of 2 treatments applied topically TID to both feet for 85 days: Clonidine Gel (3.9 mg of clonidine HCl total daily dose), or Placebo Gel (vehicle without clonidine). Approximately 140 adult subjects with symmetrical distal PDN were expected to be randomized into the study. However, a pre-planned fully blinded interim analysis was performed when 70 subjects had completed the study for the purpose of re estimating sample size. Following the recommendation of the independent, third party statistician who conducted the interim analysis, the sample size was adjusted to allow approximately 260 subjects to be randomized into the study.

The study included 5 phases: Screening Phase (up to 21 days duration), Baseline Phase (Day 14 to Day 8), Placebo Lead in Phase (Day -7 to Day 1), Double blind Treatment Phase (85 days), and a Post-treatment Follow up Phase (7 days, only for subjects not enrolling in the open label long term safety study, CLO 311).

ELIGIBILITY:
Inclusion Criteria:

* The subject has provided written informed consent.
* The subject is an outpatient aged 18 to 85 years (inclusive) at the time of the Screening Visit.
* The subject has Type 1 or Type 2 diabetes mellitus with glycemic control that has been optimized and has been stable on diet therapy, oral anti-hyperglycemic agents and/or insulin, for at least three (3) months prior to the Screening Visit.
* The subject must be a male or non-pregnant, non-lactating female. Females must be practicing an acceptable method of birth control, or be surgically sterile or postmenopausal (amenorrhea for ≥12 months). Non-pregnancy will be confirmed (as applicable) by a pregnancy test conducted at the Screening and Randomization Visits. Double-barrier methods, hormonal contraceptives, and abstinence are acceptable birth control methods for this study.
* The subject has chronic pain attributable to a symmetrical stocking distribution neuropathy in the lower extremities for at least three (3) months. A loss of distal sensation and/or tingling paresthesia primarily in the toes and fingers is acceptable, but must be of secondary importance to the distal neuropathic pain. Pain should be clearly localized to the area of neuropathy (feet) and subjects should be able to distinguish this pain (the target pain) from other painful areas and conditions.
* The subject has an average pain score relevant to the target pain in the feet of ≥4 on an 11-point Numeric Pain Rating Scale over the previous 24 hours at Screening.
* The subject has a pain score of at least 2, on the 11-point Numeric Pain Rating Scale , within 30 minutes following topical 0.1% capsaicin application with occlusive dressing to the pretibial area.
* The subject has a mean daily average pain score relevant to the target pain in the feet of ≥4 on an 11-point Numeric Pain Rating Scale during the Baseline Phase.
* The subject has met the pain evaluation and scoring criteria at the end of the Placebo Lead-in Phase by having a mean daily average pain score relevant to the target pain in the feet of ≥4 on an 11-point Numeric Pain Rating Scale without having a decrease in their pain score greater than 20% compared to the Baseline Phase score in the 11-point Numeric Pain Rating Scale .
* The subject has been medically stable for at least 30 days prior to the Screening Visit, and in the opinion of the Investigator, is in otherwise good general health based on medical history, physical examination, ECG, and laboratory evaluation.
* If taking chronic oral pain medications, the subject must be on a stable regimen for at least 14 days prior to the Baseline Visit with the expectation that the medications, dose(s) and schedule will remain stable throughout the study. For medications containing non-steroidal anti-inflammatory drugs (NSAIDs) and aspirin, subjects must be on a stable dose for at least 7 days prior to the Baseline Visit. As needed pain medications will be limited to acetaminophen from Day -8 until the end of the treatment period. Low dose aspirin (81 mg/day) is not considered as analgesic therapy.
* Subject is compliant with daily pain assessments during the Baseline Phase and Placebo Lead in Phase of the study by recording their Numeric Pain Rating Scale score at least 5 days and the last 3 days of the previous 7 days.
* Subject is alert and has the capabilities of applying topical gel to both feet three times daily. A caregiver, trained by the study staff to apply study drug, would be a suitable alternative to self-application of the treatment.

Exclusion Criteria:

* The subject has neuropathy secondary to non-diabetic causes in the opinion of the Investigator (e.g., significant vasculitis, collagen vascular disorder, familial neuropathy, alcoholism, pernicious anemia, hepatitis, malignancy, syphilis, post-herpetic neuralgia, chronic inflammatory demyelinating polyradiculopathy, human immunodeficiency virus [HIV], medication-induced neuropathy, vitamin B12 deficiency).
* The subject has a significant neurological disorder or a condition that can cause symptoms that mimic peripheral neuropathy or might confound assessment of painful diabetic neuropathy (e.g., stroke with distal neurological deficit, mononeuritis multiplex, lumbar radiculopathy, multiple sclerosis) or has significant asymmetric neuropathic signs and symptoms.
* The subject has other sustained pain with intensity at or greater than the bilateral neuropathic pain in the feet/toes.
* The subject is using an implanted medical device (e.g., spinal cord stimulator, intrathecal pump, or peripheral nerve stimulator) for the treatment of pain.
* The subject has no pin-prick sensitivity to Neuropen testing of non-calloused areas of the foot.
* The subject is clinically hypotensive with a resting diastolic blood pressure <60 mm Hg or a systolic blood pressure <90 mm Hg.
* The subject has recent history (within the past 3 months) or current symptoms of orthostatic hypotension with a sudden fall in blood pressure on standing accompanied by dizziness and lightheadedness.
* The subject has a history of foot or toe amputation, or an active foot or toe ulcer.
* The subject has any significant or unstable medical or psychiatric condition that, in the opinion of the Investigator, would interfere with his/her ability to participate in the study.
* The subject has a history of substance abuse disorder as defined by the Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) within the past year, has current evidence for substance abuse disorder, is receiving medicinal treatment for drug abuse, or tests positive upon urine drug screen for a non-prescribed substance of abuse.
* The subject has used capsaicin on the feet for greater than 2 consecutive weeks in the previous 3 months.
* The subject has symptomatic or severe coronary insufficiency, clinically significant cardiac conduction disturbances, myocardial infarction (within last 12 months), moderate to severe cerebrovascular disease, or severe chronic obstructive pulmonary disease (COPD) requiring oxygen therapy.
* The subject has a serum creatinine value >2.0 mg/dL or a value for alanine transaminase (ALT) or aspartate transaminase (AST) >2.5 times the upper limit of normal at Screening.
* The subject was dosed with an investigational drug within 30 days prior to the Screening Visit.
* The subject is likely to be noncompliant or unreliable in providing pain ratings as judged by the Investigator.
* The subject has evidence of clinically significant peripheral vascular disease as evidenced by history of intermittent claudication or evidence of vascular ulcers, including venous stasis ulcers.
* The subject has had prior treatment with clonidine topical gel.
* The subject is currently taking or has taken clonidine in any form (oral, transdermal patch) over the past 4 weeks.
* The subject has known hypersensitivity or intolerance to clonidine.
* Except for acetaminophen, the subject is currently receiving any medications that could affect neuropathic pain and is not at a stable dose for at least 14 days prior to the Baseline Visit (other than medications containing NSAIDs and aspirin which must be stable for 7 days prior to the Baseline Visit).
* The subject is receiving non-oral pain medication(s) (transdermal, topical, subcutaneous, intramuscular, intravenous, intrarectal, sublingual, transmucosal) and/or using "alternative medicine" products or techniques (acupuncture, naturopathy, homeopathy, etc.) for pain treatment ≤7 days prior to the Baseline Visit.
* Subject has a history of malignancy within the past 5 years with the exception of successfully treated non-metastatic basal cell or squamous cell carcinomas of the skin and/or localized carcinoma in situ of the cervix.
* The subject has been hospitalized within 30 days of the Screening Visit, or is planning to have surgery during the study period.
* The subject has clinical evidence of pedal edema or venous stasis disease associated with significant skin changes on physical examination.
* The subject has a clinically relevant painful foot condition, such as tarsal tunnel syndrome, plantar fasciitis, Morton's neuroma, painful bunion, or arthritis of the foot/ankle, or has a condition that may be associated with numbness in the foot.
* The subject has any dermatologic condition of the lower extremities that could affect study drug absorption (e.g., severe edema).
* The subject has current symptoms of depression with a Beck Depression Inventory -II score >19 at Screening.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2014-03; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aziz Shaibani, MD, Principal Investigator — Nerve & Muscle Center of Texas
Locations (23):
- United States (23):
  - Phoenix, Arizona
  - Santa Monica, California
  - Walnut Creek, California
  - Milford, Connecticut
  - Waterbury, Connecticut
  - Bradenton, Florida
  - Brandon, Florida
  - Jupiter, Florida
  - Miami, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Columbus, Georgia
  - Evansville, Indiana
  - Kansas City, Kansas
  - Hazelwood, Missouri
  - Winston-Salem, North Carolina
  - Warwick, Rhode Island
  - Mt. Pleasant, South Carolina
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Virginia Beach, Virginia
  - Renton, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Serednicki WT, Wrzosek A, Woron J, Garlicki J, Dobrogowski J, Jakowicka-Wordliczek J, Wordliczek J, Zajaczkowska R. Topical clonidine for neuropathic pain in adults. Cochrane Database Syst Rev. 2022 May 19;5(5):CD010967. doi: 10.1002/14651858.CD010967.pub3. PMID 35587172

RESULTS

PARTICIPANT FLOW:
Groups:
- Clonidine Gel 0.1%: Clonidine hydrochloride topical gel, 0.1%
  Clonidine Gel 0.1%
- Placebo: Placebo gel of identical appearance as active treatment
  Placebo
Period: Overall Study
Arm/Group | Clonidine Gel 0.1% | Placebo
Started | 130 | 130
Completed | 117 | 114
Not Completed | 13 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clonidine Gel 0.1% | Placebo | Total
Number analyzed (Participants) | 130 | 130 | 260
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.58 (10.458) | 59.64 (11.226) | 60.11 (10.838)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 58 | 108
  Male | 80 | 72 | 152
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 32 | 50
  Not Hispanic or Latino | 112 | 98 | 210
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 30 | 31 | 61
  White | 95 | 97 | 192
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 130 | 130 | 260

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 84 (Week 12) in Numeric Pain Rating Scale Score
Description: The Numeric Pain Rating Scale is a single reading that measures the patients interpretation of their pain on a scale from 0, no pain to 10, worst pain imaginable. The change from baseline can range from -10 to 10. The change from Baseline (averaged over Day -14 to Day -8) to End-of-Treatment (averaged over Days 78 to 84 [±3 days]) in the Numeric Pain Rating Scale score assessing the "average pain in the past 24 hours in the painful areas of the feet" averaged over Days 78 to 84 compared to the 7 days at the Baseline Phase (Days -14 to -8). For the primary efficacy endpoint, the mean change in pain intensity from Baseline to Week 12 was analyzed using an analysis of covariance (ANCOVA) model with the Baseline pain intensity score serving as a covariate. The statistical model also included treatment, site, site by treatment interaction, and strata. If the site by treatment interaction term was not significant at the 0.1 level, then it was excluded from the model.
Time Frame: The change from Baseline (averaged over Day -14 to Day -8) to End-of-Treatment (averaged over Days 78 to 84 [±3 days])
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clonidine Gel 0.1% | Placebo
Number analyzed (Participants) | 130 | 130
units on a scale | -1.6 (0.17) | -1.6 (0.19)
Statistical Analysis 1: Comparison: Clonidine Gel 0.1% vs Placebo; Test type: Superiority; p = 0.4503, Mixed Models Analysis — MMRM imputing for missing data

2. Secondary Outcome: Mean Daily Worst Pain Intensity Numeric Pain Rating Scale Scores
Description: The Numeric Pain Rating Scale is a single reading that measures the patients interpretation of their pain on a scale from 0, no pain to 10, worst pain imaginable. The change from baseline can range from -10 to 10. The change from Baseline (worst score from Day -14 to Day -8) to End-of-Treatment (worst score during Days 78 to 84 [±3 days]) in the Numeric Pain Rating Scale score assessing the "worst pain in the past 24 hours in the painful areas of the feet" from Days 78 to 84 compared to the 7 days at the Baseline Phase (Days -14 to -8). For the endpoint, the change in worst pain intensity from Baseline to Week 12 was analyzed using an analysis of covariance (ANCOVA) model with the Baseline worst pain intensity score serving as a covariate. The statistical model also included treatment, site, site by treatment interaction, and strata. If the site by treatment interaction term was not significant at the 0.1 level, then it was excluded from the model.
Time Frame: The change from Baseline (worse over Day -14 to Day -8) to End-of-Treatment (worse over Days 78 to 84 [±3 days])
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clonidine Gel 0.1% | Placebo
Number analyzed (Participants) | 130 | 130
units on a scale | -1.4 (0.11) | -1.4 (0.11)
Statistical Analysis 1: Comparison: Clonidine Gel 0.1% vs Placebo; Test type: Superiority; p = 0.7350, Mixed Models Analysis — MMRM imputing for missing data

ADVERSE EVENTS:
Arm/Group | Clonidine Gel 0.1% | Placebo
All-Cause Mortality (participants affected / at risk) | 0/130 | 0/130
Serious Adverse Events (participants affected / at risk) | 12/130 | 7/130
Other Adverse Events (participants affected / at risk) | 38/130 | 58/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clonidine Gel 0.1% (N=130) | Placebo (N=130)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic cardiomyophathy (Cardiac disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophagitits (Gastrointestinal disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Electrocardiogram t wave inversion (Investigations) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Arterial stenosis (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clonidine Gel 0.1% (N=130) | Placebo (N=130)
Back pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 11 (11)
Pain in extrimity (Musculoskeletal and connective tissue disorders) | 2 (2) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 7 (7)
Heachache (Nervous system disorders) | 10 (10) | 20 (20)
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (3) | 8 (8)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 7 (7) | 1 (1)
Oedema peripheral (General disorders) | 7 (7) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days